CLINICAL TRIAL: NCT06933953
Title: Psychometric Validation of the Foot Health Status Questionnaire in French Language
Brief Title: Validation of the Foot Health Status Questionnaire in French Language
Acronym: FHSQ-Fr
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUO-2024-12
Record Dates: First submitted 2024-12-16; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Patients With Foot Problems
Keywords: Surveys and Questionnaires; FHSQ French translation; Health status; Foot; Validity; Reliability
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with foot problems (Other): Patients will complete many questionnaires : FHSQ-fr, Foot Function Index, EQ-5D-5L, Visual Analog Pain Scale, SF-12
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients will complete various questionnaires at J0: FHSQ-Fr, EQ-5D-5L, Foot Function Index, Visual analog pain scale, SF-12.
  Patients who needs to come back for a visit at Day 7 (+ 3 days) will complete the FHSQ-Fr questionnaire for a second time

SUMMARY:
A French foot health survey showed that 73% of people examined felt pain and 38% don't left their home, which suggest a reduction in their life's quality and autonomy. Developed by Paul Bennett, FHSQ is a foot health-specific self administrated questionnaire. It sensitively detects changes in patients' foot health status, whatever their pathology, across multidimensional concepts of their quality of life. Actually, more than 150 scientific publications have cited it. Reliable and valid, it has already been translated and validated in multiple languages, but not in French. The subject of this study is to validate the translated and cross-cultural adapted French version FHSQ-fr through its psychometric results of validity and reliability. The study follows a 2-stage methodology.

The first, already completed, consisted of (back)translating the Australian FHSQ questionnaire into French by a scientific committee in order to obtain a pre-final version.

The second is to validate this final version using appropriate statistical analysis, including correlations studies with other French validated questionnaires, to determine its psychometric characteristics.

DETAILED DESCRIPTION:
To assess validity, 150 volunteers will fill out French validated questionnaires, Foot Function Index (FFI), EuroQuality of life 5D-5L (EQ5D) , Visual Analogic Pain Scale (VAPS), and Short Form 12 Health survey (SF12). They will be evaluated about their pain, morphology, function and posture of their feet as usual at a podiatric school. To assess reliability, 50 respondents from the 150 who didn't receive any treatment after 7 to 10 days, will complete the FHSQ-fr again. It would improve knowledge of the status of foot health and its related quality of life in the general population and those suffering from specific pathologies such as diabetes or rheumatoid arthritis, the effectiveness of certain treatments on the same foot condition, and their evolutions using longitudinal studies in France. At the international, the French future results of studies using this clinimetric tool could be compared with those who come from other countries, and integrated to the Australian author's " Bigdataset" which compares, analyses and predicts more accurately the clinically significant efficacy of a treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients coming to IFRES in Alençon (61) France for a pedicure or podiatry appointment,
2. Age >= 18
3. knowing how to speak, read and write French.

Exclusion Criteria:

1. Have already taking part in this research before the proposition to get in.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Internal consistency | Day 0
  It is evaluated using Cronbach's alpha coefficient "α", which measures the internal consistency of a set of items, scales or sub-scales for a single clinical dimension. The value of this index is less than or equal to 1, and the closer alpha is to 1, the stronger it is. α" > 0.7 or >0.8 is considered fairly high. However, the coefficient must not be too close to 1, otherwise the items are redundant and duplicate each other.
Temporal stability of patients' questionnaire scores FHSQ-en V 1.02 | Day 0 and day 7
  It is measured by the Intraclass Correlation Coefficient (ICC) and its 95% confidence interval, and/or the Pearson Correlation Coefficient.
  By convention, fidelity is said to be:
  * Very good if ICC ≥0 91
  * Good if 0.9 ≤ ICC ≤ 0.71
  * Moderate if 0.70 ≤ ICC ≤ 0.51
  * Poor if 0.5 ≤ ICC ≤ 0.31
  * Very poor or nil if ICC ≤ 0.3
Measurement error | Day 0
  To apply the criterion of good measurement error, the MIC (Minimal Important Change), the SDC (Smallest Detectable Change) or the LoA (Limits of Agreement) load will be calculated using a longitudinal approach based on anchoring.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine GUYET, Principal Investigator — IFRES of Alençon
Locations (1):
- Ifres Ecole de Pedicure Podologie, Alençon, France

REFERENCES:
- [Background] Burzykowski T, Molenberghs G, Abeck D, Haneke E, Hay R, Katsambas A, Roseeuw D, van de Kerkhof P, van Aelst R, Marynissen G. High prevalence of foot diseases in Europe: results of the Achilles Project. Mycoses. 2003 Dec;46(11-12):496-505. doi: 10.1046/j.0933-7407.2003.00933.x. PMID 14641624
- [Background] Lopez-Lopez D, Perez-Rios M, Ruano-Ravina A, Losa-Iglesias ME, Becerro-de-Bengoa-Vallejo R, Romero-Morales C, Calvo-Lobo C, Navarro-Flores E. Impact of quality of life related to foot problems: a case-control study. Sci Rep. 2021 Jul 15;11(1):14515. doi: 10.1038/s41598-021-93902-5. PMID 34267276
- [Background] Valensi P, Girod I, Baron F, Moreau-Defarges T, Guillon P. Quality of life and clinical correlates in patients with diabetic foot ulcers. Diabetes Metab. 2005 Jun;31(3 Pt 1):263-71. doi: 10.1016/s1262-3636(07)70193-3. PMID 16142017
- [Background] Bennett PJ, Patterson C, Wearing S, Baglioni T. Development and validation of a questionnaire designed to measure foot-health status. J Am Podiatr Med Assoc. 1998 Sep;88(9):419-28. doi: 10.7547/87507315-88-9-419. PMID 9770933
- See also: A few figures on foot health in France - UFSP — https://www.sante-du-pied.org/lufsp/les-chiffres/